CLINICAL TRIAL: NCT02672683
Title: Non Invasive Detection of Acute Rejection by Circulating microRNAs in Cardiac Transplantation: a Multicenter Prospective Study
Brief Title: Non Invasive Detection of Cardiac Allograft Rejection by Circulating microRNAs
Acronym: MIRRACLE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: AOR 14086
Record Dates: First submitted 2015-11-30; First posted 2016-02-03 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cardiac Transplantation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate the level of expression of 4 circulating microRNAs in the serum using RT-PCR. A pilote study with cardiac transplant patients has shown that expression of these microRNAs could discriminate patients with a histologically proven rejection from patient displaying a normal endomyocardial biopsy. The signature must be confirmed in unselected patients and its stability evaluated according to clinical, biological and immunological parameters of included patients.

DETAILED DESCRIPTION:
Heart transplantation is the only available long-term treatment option for patients with terminal heart failure.

Despite considerable progress in immunosuppressive regimens, allograft rejection remains a major cause of graft loss.

Majority of cardiac allograft rejection are asymptomatic. Only severe rejection goes along with cardiac dysfunction. This clinical latency makes the cardiac rejection diagnostic difficult and has ruled modalities of detection of cardiac rejection.

The cornerstone of rejection diagnosis and post-transplant follow-up relies on endomyocardial biopsy (EMB) and classical histopathology assessment. Echocardiography and MRI are neither sensitive nor specific enough to replace EMB. Majority of transplant centers thus evaluate rejection using iterative protocol biopsies. These cardiac allograft monitoring protocols are heavy, with 15 to 20 EMB in the first year of transplantation and 1 to 2 EMB each year after the first year. EMB are invasive procedure with a low but not zero risk of severe adverse events. Repetition of EMB is associated with tricuspid regurgitation due to valvular complications. Moreover incidence of cardiac rejection explains the cost-effectiveness of EMBs: 50 to 70% of biopsies are normal.

The goal is thus to detect rejection in the blood by measuring expression levels of 4 circulating microRNAs in patients' sera by RT-PCR. The seric expression levels of these 4 circulating microRNAs will be compared to the histopathological diagnosis made on concomitant endomyocardial biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cardiac transplant at the time of inclusion
* Patients transplanted for less than 10 years and having an annual follow-up
* Patients with a biopsy evaluation during their follow-up, at month 1, 3, 6, 12 (newly transplanted) and annually (newly and already transplanted patients) and concomitant routine blood work
* Patients not opposed to the study
* Patients with assessment of anti-donor specific antibodies during the study period

Exclusion Criteria:

* Patients with a multi-organ transplantation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with a cardiac transplant
Sampling Method: Non-Probability Sample
Enrollment: 461 (Actual)
Dates: Start 2016-09-26 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2019-03-26 (Actual)

PRIMARY OUTCOMES:
Comparison of circulating MicroRNAs measurement in serum with histopathological diagnosis of rejection on concomitant endomyocardial biopsy | one month
Comparison of circulating MicroRNAs measurement in serum with histopathological diagnosis of rejection on concomitant endomyocardial biopsy | 3 months
Comparison of circulating MicroRNAs measurement in serum with histopathological diagnosis of rejection on concomitant endomyocardial biopsy | 6 months
Comparison of circulating MicroRNAs measurement in serum with histopathological diagnosis of rejection on concomitant endomyocardial biopsy | 12 months

SECONDARY OUTCOMES:
Comparison of circulating MicroRNAs measurement in serum with histopathological diagnosis of rejection on concomitant endomyocardial biopsy | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Jean-paul Duong Van Huyen, MD, PhD, Principal Investigator — Necker Hospital, AP-HP
Locations (1):
- PARCC/ INSERM U970, Team 4, Xavier Jouven, Cardiovascular epidemiology and sudden death, Georges Pompidou European Hospital,, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Duong Van Huyen JP, Tible M, Gay A, Guillemain R, Aubert O, Varnous S, Iserin F, Rouvier P, Francois A, Vernerey D, Loyer X, Leprince P, Empana JP, Bruneval P, Loupy A, Jouven X. MicroRNAs as non-invasive biomarkers of heart transplant rejection. Eur Heart J. 2014 Dec 1;35(45):3194-202. doi: 10.1093/eurheartj/ehu346. Epub 2014 Aug 31. PMID 25176944
- [Result] Coutance G, Racape M, Baudry G, Lecuyer L, Roubille F, Blanchart K, Epailly E, Vermes E, Pattier S, Boignard A, Gay A, Bruneval P, Jouven X, Duong Van Huyen JP, Loupy A. Validation of the clinical utility of microRNA as noninvasive biomarkers of cardiac allograft rejection: A prospective longitudinal multicenter study. J Heart Lung Transplant. 2023 Nov;42(11):1505-1509. doi: 10.1016/j.healun.2023.07.010. Epub 2023 Jul 23. PMID 37487804